CLINICAL TRIAL: NCT02938585
Title: Efficacy and Safety of Turoctocog Alfa for Prophylaxis and Treatment of Bleeding Episodes in Previously Treated Chinese Patients With Haemophilia A
Acronym: guardian TM 7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-4028; U1111-1150-0765 (Other: WHO); CTR20160811 (Other: CFDA); 2013-004791-35 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic treatment (Experimental)
  Interventions: Drug: turoctocog alfa
- On-demand treatment (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — The preventative treatment is administered intravenously (i.v.) at specific intervals either every second day or three times a week. Bleeding treatment will be administered if a bleed should occur.
  Arms: Prophylactic treatment
Drug: turoctocog alfa — Treatment is administered intravenously (i.v.) during bleeds and occasionally as a preventative treatment (e.g. before physical activity)
  Arms: On-demand treatment

SUMMARY:
This trial is conducted in China. The aim of this trial is to evaluate the clinical efficacy of turoctocog alfa in treatment of bleeding episodes in Chinese patients with severe haemophilia A (FVIII≤1%).

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Age from 0 years
* With the diagnosis of severe congenital haemophilia A (FVIII≤1%)
* History of exposure days (ED) to any FVIII products fulfilling the criteria of previously treated patients:
* Patients of 12 years or above: 100 exposures days (ED) or more
* Patients below 12 years: 50 exposure days (ED) or more

Exclusion Criteria:

* Inhibitors to factor VIII (≥0.6 BU) at screening as assessed by central laboratory
* Known history of FVIII inhibitors

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chonqqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Guiyang, Guizhou
  - Novo Nordisk Investigational Site, Wuhan, Hubei
  - Novo Nordisk Investigational Site, Xining, Qinghai
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Kunming, Yunnan
  - Novo Nordisk Investigational Site, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 10 sites in mainland China.
Pre-assignment Details: Study design: This was an open-label and non-randomised trial. Participants with severe haemophilia A were administered a prophylaxis (preventive) or on-demand regimen of turoctocog alfa (trial product) at the investigator's discretion.
Groups:
- Small Children (0 to <6 Years): Participants were to receive turoctocog alfa intravenous (i.v.) injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 30 IU/kg. Prophylaxis doses ranged from 25-50 IU/kg (once every-second-day), or 25-60 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the World Federation of Haemophilia (WFH) guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their coagulation factor VIII (FVIII) activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
- Older Children (6 to <12 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 30 IU/kg. Prophylaxis doses ranged from 25-50 IU/kg (once every-second-day), or 25-60 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance, and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
- Adolescents (12 to <18 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 25 IU/kg. Prophylaxis doses ranged from 20-40 IU/kg (once every-second-day), or 20-50 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
- Adults (>=18 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. Participants who completed 6 months of treatment (prophylaxis or on-demand) in the main phase, were to continue the same treatment for up to approximately 18 months (extension phase). Participants were allowed to switch between treatments in the 'extension phase'. The recommended prophylaxis starting dose was 25 IU/kg. Prophylaxis doses ranged from 20-40 IU/kg (once every-second-day), or 20-50 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
Period: Overall Study
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Started | 9 | 33 | 11 | 15
Exposed to Prophylaxis Regimen (As participants were allowed to change regimen in EXT phase, some participants were exposed to both) | 9 | 31 | 11 | 12
Exposed to On-demand Regimen (As participants were allowed to change regimen in EXT phase, some participants were exposed to both) | 1 | 7 | 1 | 8
Completed | 9 | 32 | 11 | 10
Not Completed | 0 | 1 | 0 | 5
Not completed — Withdrawal by parent or guardian | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set, which included all dosed participants with data after dosing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years) | Total
Number analyzed (Participants) | 9 | 33 | 11 | 15 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.00 (1.12) | 8.70 (1.91) | 14.55 (1.92) | 31.00 (11.20) | 13.94 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 9 | 33 | 11 | 15 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 33 | 11 | 15 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 33 | 11 | 15 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Haemostatic Effect of Turoctocog Alfa (Treatment of Bleeds): 6 Months
Description: The haemostatic effect of turoctocog alfa when used for treatment of bleeding episodes in both prophylaxis and on-demand regimen was evaluated during month 0-6. The effect was assessed on a four-point scale for haemostatic response, excellent, good, moderate and none.
Time Frame: Month 0-6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants with bleeding episodes, from both prophylaxis and on-demand regimen.
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Groups:
- Adults (>=18 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 25 IU/kg. Prophylaxis doses ranged from 20-40 IU/kg (once every-second-day), or 20-50 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 6 | 20 | 6 | 15
Number analyzed (Bleeding episodes) | 48 | 245 | 28 | 290
Bleeding episodes
  Excellent | 35 | 156 | 20 | 190
  Good | 12 | 73 | 8 | 87
  Moderate | 1 | 15 | 0 | 13
  None | 0 | 0 | 0 | 0
  Missing | 0 | 1 | 0 | 0

2. Secondary Outcome: Haemostatic Effect of Turoctocog Alfa (Treatment of Bleeds): 24 Months
Description: The haemostatic effect of turoctocog alfa when used for treatment of bleeding episodes in both prophylaxis and on-demand regimen was evaluated during month 0-24. The effect was assessed on a four-point scale for haemostatic response, excellent, good, moderate and none.
Time Frame: Month 0-24
Population: as for outcome 1
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: Bleeding episodes
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 7 | 24 | 8 | 15
Number analyzed (Bleeding episodes) | 65 | 405 | 53 | 402
Bleeding episodes
  Excellent | 45 | 275 | 42 | 272
  Good | 18 | 103 | 11 | 116
  Moderate | 2 | 26 | 0 | 14
  None | 0 | 0 | 0 | 0
  Missing | 0 | 1 | 0 | 0

3. Secondary Outcome: Incidence Rate of Inhibitory Antibodies Against FVIII (≥0.6 BU): 6 Months
Description: This endpoint presented 'percentage of participants with inhibitory antibodies against FVIII (≥0.6 BU)' in both prophylaxis and on-demand regimen, evaluated during month 0-6.
Time Frame: Month 0-6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants, from both prophylaxis and on-demand regimen.
Measure: Number; unit: Percentage of participants
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
Percentage of participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence Rate of Inhibitory Antibodies Against FVIII (≥0.6 BU): 24 Months
Description: This endpoint presented 'percentage of participants with inhibitory antibodies against FVIII (≥0.6 BU)' in both prophylaxis and on-demand regimen, evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
Percentage of participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Bleeds (Total Bleeds Assessed as Annual Bleeding Rate) Per Participant: 6 Months
Description: Number of bleeds (total bleeds assessed as annual bleeding rate) per participant in the prophylaxis regimen was evaluated during month 0-6. The annualised bleeding rate was analysed by a negative binomial model.
Time Frame: Month 0-6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants from the prophylaxis regimen.
Measure: Number (95% Confidence Interval); unit: Bleeding episodes/year
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 8 | 26 | 10 | 7
Bleeding episodes/year | 4.36 [1.71 to 11.14] | 4.11 [2.15 to 7.87] | 2.34 [0.81 to 6.72] | 10.67 [5.53 to 20.57]

6. Secondary Outcome: Number of Bleeds (Total Bleeds Assessed as Annual Bleeding Rate) Per Participant: 24 Months
Description: Number of bleeds (total bleeds assessed as annual bleeding rate) per participant in the prophylaxis regimen was evaluated during month 0-24. The annualised bleeding rate was analysed by a negative binomial model.
Time Frame: Month 0-24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Bleeding episodes/year
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 31 | 11 | 12
Bleeding episodes/year | 2.28 [1.02 to 5.10] | 2.63 [1.53 to 4.51] | 1.97 [0.83 to 4.67] | 4.97 [1.96 to 12.60]

7. Secondary Outcome: Consumption of Turoctocog Alfa for Bleeding Treatment: Average Dose to Treat a Bleed (6 Months)
Description: Average dose of turoctocog alfa used to treat a bleed in both prophylaxis and on-demand regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg BW
Units Other Than Participants: doses
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 6 | 20 | 6 | 15
Number analyzed (doses) | 69 | 361 | 60 | 400
IU/kg BW | 42.96 (5.35) | 36.69 (14.04) | 46.79 (5.31) | 20.29 (6.48)

8. Secondary Outcome: Consumption of Turoctocog Alfa for Bleeding Treatment: Average Dose to Treat a Bleed (24 Months)
Description: Average dose of turoctocog alfa used to treat a bleed in both prophylaxis and on-demand regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg BW
Units Other Than Participants: doses
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 7 | 24 | 8 | 15
Number analyzed (doses) | 94 | 624 | 95 | 565
IU/kg BW | 43.99 (6.95) | 36.00 (12.32) | 43.58 (6.93) | 21.07 (7.49)

9. Secondary Outcome: Consumption of Turoctocog Alfa for Bleeding Treatment: Number of Injections Per Bleed (6 Months)
Description: Number of turoctocog alfa injections consumed to treat a bleeding episode in both prophylaxis and on-demand regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Injections
Units Other Than Participants: bleeding episodes
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 6 | 20 | 6 | 15
Number analyzed (bleeding episodes) | 48 | 245 | 28 | 290
Injections | 1.31 (0.59) | 1.22 (0.61) | 1.07 (0.26) | 1.29 (0.89)

10. Secondary Outcome: Consumption of Turoctocog Alfa for Bleeding Treatment: Number of Injections Per Bleed (24 Months)
Description: Number of turoctocog alfa injections consumed to treat a bleeding episode in both prophylaxis and on-demand regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Injections
Units Other Than Participants: bleeding episodes
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 7 | 24 | 8 | 15
Number analyzed (bleeding episodes) | 65 | 405 | 53 | 402
Injections | 1.34 (0.62) | 1.30 (0.88) | 1.09 (0.30) | 1.33 (1.21)

11. Secondary Outcome: Consumption of Turoctocog Alfa for Bleeding Treatment: IU/kg Per Bleed (6 Months)
Description: Consumption of turoctocog alfa IU/kg BW per bleed in both prophylaxis and on-demand regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg BW
Units Other Than Participants: bleeding episodes
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 6 | 20 | 6 | 15
Number analyzed (bleeding episodes) | 48 | 245 | 28 | 290
IU/kg BW | 56.60 (25.32) | 42.37 (26.54) | 48.82 (15.05) | 26.20 (17.55)

12. Secondary Outcome: Consumption of Turoctocog Alfa for Bleeding Treatment: IU/kg Per Bleed (24 Months)
Description: Consumption of turoctocog alfa IU/kg BW per bleed in both prophylaxis and on-demand regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg BW
Units Other Than Participants: bleeding episodes
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 7 | 24 | 8 | 15
Number analyzed (bleeding episodes) | 65 | 405 | 53 | 402
IU/kg BW | 59.01 (28.61) | 44.75 (34.15) | 45.07 (15.33) | 27.44 (22.52)

13. Secondary Outcome: Consumption of Turoctocog Alfa During Preventive Treatment Per Participant: Average Preventive Dose (6 Months)
Description: Average preventive dose of turoctocog alfa consumed per participant in the prophylaxis regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg BW
Units Other Than Participants: doses
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 8 | 26 | 10 | 7
Number analyzed (doses) | 530 | 1689 | 661 | 484
IU/kg BW | 47.05 (9.21) | 39.46 (7.12) | 35.40 (7.41) | 37.28 (5.22)

14. Secondary Outcome: Consumption of Turoctocog Alfa During Preventive Treatment Per Participant: Average Preventive Dose (24 Months)
Description: Average preventive dose of turoctocog alfa consumed per participant in the prophylaxis regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg BW
Units Other Than Participants: doses
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 31 | 11 | 12
Number analyzed (doses) | 2314 | 6729 | 2794 | 1999
IU/kg BW | 47.97 (8.00) | 40.33 (7.05) | 36.20 (7.15) | 38.13 (7.51)

15. Secondary Outcome: Consumption of Turoctocog Alfa During Preventive Treatment Per Participant: IU/kg Per Month (6 Months)
Description: Preventive dose of turoctocog alfa (IU/kg body weight (BW) per month) per participant in the prophylaxis regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg BW/month/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 8 | 26 | 10 | 7
IU/kg BW/month/participant | 600.3 (112.6) | 522.5 (87.59) | 454.5 (92.79) | 500.7 (84.39)

16. Secondary Outcome: Consumption of Turoctocog Alfa During Preventive Treatment Per Participant: IU/kg Per Month (24 Months)
Description: Preventive dose of turoctocog alfa (IU/kg body weight (BW) per month) per participant in the prophylaxis regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg BW/month/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 31 | 11 | 12
IU/kg BW/month/participant | 606.3 (118.5) | 533.0 (82.90) | 467.6 (91.40) | 490.8 (115.7)

17. Secondary Outcome: Consumption of Turoctocog Alfa During Preventive Treatment Per Participant: IU/kg Per Year (6 Months)
Description: Preventive dose of turoctocog alfa (IU/kg body weight per year) per participant in the prophylaxis regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg BW/year/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 8 | 26 | 10 | 7
IU/kg BW/year/participant | 7204 (1351) | 6270 (1051) | 5454 (1113) | 6009 (1013)

18. Secondary Outcome: Consumption of Turoctocog Alfa During Preventive Treatment Per Participant: IU/kg Per Year (24 Months)
Description: Preventive dose of turoctocog alfa (IU/kg body weight (BW) per year) per participant in the prophylaxis regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU/kg BW/year/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 31 | 11 | 12
IU/kg BW/year/participant | 7276 (1422) | 6396 (994.7) | 5611 (1097) | 5890 (1388)

19. Secondary Outcome: Total Consumption of Turoctocog Alfa Per Participant: IU/kg Per Month (6 Months)
Description: Total consumption of turoctocog alfa (IU/kg body weight per month) per participant in both prophylaxis and on-demand regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants from both prophylaxis and on-demand regimen.
Measure: Mean (Standard Deviation); unit: IU/kg BW/month/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
IU/kg BW/month/participant | 603.5 (141.2) | 496.0 (146.7) | 479.6 (103.9) | 377.2 (218.9)

20. Secondary Outcome: Total Consumption of Turoctocog Alfa Per Participant: IU/kg Per Month (24 Months)
Description: Total consumption of turoctocog alfa (IU/kg body weight per month) per participant in both prophylaxis and on-demand regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/kg BW/month/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
IU/kg BW/month/participant | 615.3 (123.8) | 516.7 (121.1) | 477.0 (94.37) | 429.1 (192.7)

21. Secondary Outcome: Total Consumption of Turoctocog Alfa Per Participant: IU/kg Per Year (6 Months)
Description: Total consumption of turoctocog alfa (IU/kg body weight per year) per participant in both prophylaxis and on-demand regimen was evaluated during month 0-6.
Time Frame: Month 0-6
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/kg BW/year/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
IU/kg BW/year/participant | 7242 (1695) | 5951 (1760) | 5756 (1247) | 4527 (2627)

22. Secondary Outcome: Total Consumption of Turoctocog Alfa Per Participant: IU/kg Per Year (24 Months)
Description: Total consumption of turoctocog alfa (IU/kg body weight per year) per participant in both prophylaxis and on-demand regimen was evaluated during month 0-24.
Time Frame: Month 0-24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/kg BW/year/participant
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
IU/kg BW/year/participant | 7384 (1486) | 6201 (1453) | 5724 (1132) | 5149 (2312)

23. Secondary Outcome: Frequency of Adverse Events (6 Months)
Description: Frequency of adverse events (AEs) are presented as rate of events, which was calculated as the number of AEs per patient years. All presented AEs are treatment emergent (TEAEs), which were defined as the events reported after trial product administration until the end of the post-treatment follow-up period.
Time Frame: Month 0-6
Population: The safety analysis set included participants who received at least one dose of the trial product. "Overall Number of Participants Analyzed" = number of participants from both prophylaxis and on-demand regimen.
Measure: Number; unit: Events per person-year
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
Events per person-year | 4.908 | 2.093 | 2.325 | 1.922

24. Secondary Outcome: Frequency of Adverse Events (24 Months)
Description: as for outcome 23
Time Frame: Month 0-24
Population: as for outcome 23
Measure: Number; unit: Events per person-year
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
Events per person-year | 2.941 | 1.210 | 1.074 | 1.123

25. Secondary Outcome: Frequency of Serious Adverse Events (6 Months)
Description: Frequency of serious adverse events (SAEs) are presented as rate of events, which was calculated as the number of SAEs per patient years. All presented SAEs are treatment emergent, which were defined as the events reported after trial product administration until the end of the post-treatment follow-up period.
Time Frame: Month 0-6
Population: as for outcome 23
Measure: Number; unit: Events per person-year
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
Events per person-year | 0 | 0 | 0.634 | 0

26. Secondary Outcome: Frequency of Serious Adverse Events (24 Months)
Description: as for outcome 25
Time Frame: Month 0-24
Population: as for outcome 23
Measure: Number; unit: Events per person-year
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 9 | 33 | 11 | 15
Events per person-year | 0.065 | 0 | 0.161 | 0

27. Secondary Outcome: Haemostatic Effect of Turoctocog Alfa (Surgery): 6 Months
Description: The haemostatic effect of turoctocog alfa when used for surgery was evaluated during month 0-6. The effect was assessed on a four-point scale for haemostatic response (excellent, good, moderate and none) and assessed by the investigator/surgeon on the day of surgery (day 1) and on the last day in the post-operative period the participant was at the trial/surgery site.
Time Frame: Month 0-6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants who underwent surgeries, from both prophylaxis and on-demand regimen.
Measure: Number; unit: Surgeries
Units Other Than Participants: surgeries
Groups:
- Minor Surgery: Participants who underwent minor surgery (including tooth extraction) during month 0-6 (main phase), were treated with turoctocog alfa according to WFH recommendations and were to maintain FVIII activity levels at 30-60 IU/dL. Minor surgery: Any invasive operative procedure in which only skin, mucous membranes, or superficial connective tissue was manipulated. Examples of minor surgery: vascular cutdown for catheter/fistula placement, implanting pumps or central venous access device (CVAD) in subcutaneous tissue, biopsies or placement of probes, leads, or catheters requiring the entry into a body cavity only through a needle/guidewire.
- Major Surgery: Participants who underwent major surgery during month 0-6 (main phase), were treated with turoctocog alfa according to WFH recommendations and were to maintain FVIII activity levels at 80-100 IU/dL pre- and postoperatively. Major surgery: Any invasive operative procedure where any one or more of the following occurred: 1) A body cavity was entered. 2) A mesenchymal barrier (e.g. pleura, peritoneum or dura) was crossed. 3) A fascial plane was opened. 4) An organ was removed. 5) Normal anatomy was operatively altered.
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 3 | 3
Number analyzed (surgeries) | 3 | 3
Surgeries
  During surgery: Excellent | 2 | 1
  During surgery: Good | 1 | 2
  During surgery: Moderate | 0 | 0
  During surgery: None | 0 | 0
  After surgery: Excellent | 3 | 2
  After surgery: Good | 0 | 1
  After surgery: Moderate | 0 | 0
  After surgery: None | 0 | 0

28. Secondary Outcome: Haemostatic Effect of Turoctocog Alfa (Surgery): 24 Months
Description: The haemostatic effect of turoctocog alfa when used for surgery was evaluated during month 0-24. The effect was assessed on a four-point scale for haemostatic response (excellent, good, moderate and none) and assessed by the investigator/surgeon on the day of surgery (day 1) and on the last day in the post-operative period the participant was at the trial/surgery site. Haemostatic response of 'not applicable' indicated that turoctocog alfa was not used.
Time Frame: Month 0-24
Population: as for outcome 27
Measure: Number; unit: Surgeries
Units Other Than Participants: surgeries
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 5 | 3
Number analyzed (surgeries) | 6 | 4
Surgeries
  During surgery: Excellent | 3 | 1
  During surgery: Good | 1 | 3
  During surgery: Moderate | 0 | 0
  During surgery: None | 0 | 0
  During surgery: Not applicable | 2 | 0
  After surgery: Excellent | 5 | 2
  After surgery: Good | 0 | 2
  After surgery: Moderate | 0 | 0
  After surgery: None | 0 | 0
  After surgery: Not applicable | 1 | 0

29. Secondary Outcome: Loss of Blood (Surgery): 6 Months
Description: Loss of blood was evaluated during month 0-6: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant was at the trial/surgery site whatever comes first.
Time Frame: Month 0-6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants who underwent surgeries, from both prophylaxis and on-demand regimen. "Overall Number of Units Analyzed" = number of surgeries where blood loss happened.
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgeries with blood loss
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 3 | 3
Number analyzed (surgeries with blood loss) | 2 | 3
mL | 2.0 (1.4) | 106.7 (90.2)

30. Secondary Outcome: Loss of Blood (Surgery): 24 Months
Description: Loss of blood was evaluated during month 0-24: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant was at the trial/surgery site whatever comes first.
Time Frame: Month 0-24
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: surgeries with blood loss
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 5 | 3
Number analyzed (surgeries with blood loss) | 2 | 4
mL | 2.0 (1.4) | 81.3 (89.5)

31. Secondary Outcome: Requirements for Transfusion (Surgery): 6 Months
Description: Surgeries required transfusion was evaluated during month 0-6: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant was at the trial/surgery site whatever comes first.
Time Frame: Month 0-6
Population: as for outcome 27
Measure: Number; unit: Surgeries
Units Other Than Participants: surgeries
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 3 | 3
Number analyzed (surgeries) | 3 | 3
Surgeries | 0 | 0

32. Secondary Outcome: Requirements for Transfusion (Surgery): 24 Months
Description: Surgeries required transfusion was evaluated during month 0-24: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant was at the trial/surgery site whatever comes first.
Time Frame: Month 0-24
Population: as for outcome 27
Measure: Number; unit: Surgeries
Units Other Than Participants: surgeries
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 5 | 3
Number analyzed (surgeries) | 6 | 4
Surgeries | 0 | 0

33. Secondary Outcome: Adverse Events (Surgery): 6 Months
Description: TEAEs during surgery were recorded during month 0-6: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant was at the trial/surgery site whatever comes first. TEAEs were defined as the events reported after trial product administration until the end of the post-treatment follow-up period.
Time Frame: Month 0-6
Population: The safety analysis set included participants who received at least one dose of the trial product. "Overall Number of Participants Analyzed" = number of participants who underwent surgeries, from both prophylaxis and on-demand regimen.
Measure: Number; unit: Events
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 3 | 3
Events | 1 | 1

34. Secondary Outcome: Adverse Events (Surgery): 24 Months
Description: TEAEs during surgery were recorded during month 0-24: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant was at the trial/surgery site whatever comes first. TEAEs were defined as the events reported after trial product administration until the end of the post-treatment follow-up period.
Time Frame: Month 0-24
Population: as for outcome 33
Measure: Number; unit: Events
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 5 | 3
Events | 4 | 1

35. Secondary Outcome: Serious Adverse Events (Surgery): 6 Months
Description: Treatment emergent serious adverse events occurred during surgery were recorded from month 0 to month 6: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant is at the trial/surgery site whatever comes first. Treatment emergent events were defined as the events reported after trial product administration until the end of the post-treatment follow-up period.
Time Frame: Month 0-6
Population: as for outcome 33
Measure: Number; unit: Events
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 3 | 3
Events | 0 | 0

36. Secondary Outcome: Serious Adverse Events (Surgery): 24 Months
Description: Treatment emergent serious adverse events occurred during surgery were recorded from month 0 to month 24: on the day of surgery (day 1) and during the post-operative period days 2-7 or until the last day the participant is at the trial/surgery site whatever comes first. Treatment emergent events were defined as the events reported after trial product administration until the end of the post-treatment follow-up period.
Time Frame: Month 0-24
Population: as for outcome 33
Measure: Number; unit: Events
Arm/Group | Minor Surgery | Major Surgery
Number analyzed (Participants) | 5 | 3
Events | 0 | 0

37. Secondary Outcome: Change in Total Scores for Reported Health-related Quality of Life (for Participants): Month 6
Description: Reported results are baseline (month 0) and change from baseline (at month 6) of end of disease and age specific HRQOL. HRQOL was collected through use of the patient reported outcome (PRO) instruments, HAEMO-QOL (for children (8-12 years)/adolescents (13-16 years)) and HAEM-A-QOL (for adults (>=17 years)). HAEMO-QOL assessment included questions on physical health, feeling, view of yourself, family, friends, perceived support, other persons, sports and school, dealing with haemophilia, treatment, future, and relationships. HAEM-A-QOL assessment included questions on physical health, feeling, view of yourself, sports and leisure, work and school, dealing with haemophilia, treatment, future, family planning, and partnership and sexuality. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Observed mean of the means of all the questions for HAEMO-QOL and HAEM-A-QOL, respectively are presented.
Time Frame: Month 0, Month 6
Population: The full analysis set included all dosed participants with data after dosing. "Overall Number of Participants Analyzed" = number of participants from both prophylaxis and on-demand regimen. "Number Analyzed" = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Scores
Groups:
- Older Children (8 to 12 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 30 IU/kg (for <12 years participants) and 25 IU/kg (for 12 years participants). Prophylaxis doses ranged from 25-50 IU/kg (for <12 years participants) and 20-40 IU/kg (for 12 years participants) with every-second-day treatment, or 25-60 IU/kg (for <12 years participants) and 20-50 IU/kg (for 12 years participants) with 3-times-weekly treatment. Bleeds and surgeries were treated in the same way as for the other two treatment groups (adolescents (13 to 16 years) and adults (17 and older)).
- Adults (17 and Older): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 25 IU/kg. Prophylaxis doses ranged from 20-40 IU/kg (once every-second-day), or 20-50 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
Arm/Group | Older Children (8 to 12 Years) | Adolescents (12 to <18 Years) | Adults (17 and Older)
Number analyzed (Participants) | 22 | 6 | 18
Scores
  Baseline | 41.3 (16.4) | 42.2 (12.8) | 47.2 (13.8)
  Change from baseline | -6.8 (14.5) | -3.5 (3.6) | -3.4 (12.8)

38. Secondary Outcome: Change in Total Scores for Reported Health-related Quality of Life (for Participants): Month 24
Description: Reported results are baseline (month 0) and change from baseline (at month 24) of end of disease and age specific HRQOL. HRQOL was collected through use of the patient reported outcome (PRO) instruments, HAEM-A-QOL (for adults (>=17 years)) and HAEMO-QOL (for children (8-12 years)/adolescents (13-16 years)). HAEM-A-QOL assessment included questions on physical health, feeling, view of yourself, sports and leisure, work and school, dealing with haemophilia, treatment, future, family planning, and partnership and sexuality. HAEMO-QOL assessment included questions on physical health, feeling, view of yourself, family, friends, perceived support, other persons, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Observed mean of the means of all the questions for HAEM-A-QOL and HAEMO-QOL, respectively are presented.
Time Frame: Month 0, Month 24
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Scores
Groups:
- Older Children (8 to 12 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. Participants who completed 6 months of treatment (prophylaxis or on-demand) in the main phase, were to continue the same treatment for up to approximately 18 months (extension phase). Participants were allowed to switch between treatments in the 'extension phase'. The recommended prophylaxis starting dose was 30 IU/kg (for <12 years participants) and 25 IU/kg (for 12 years participants). Prophylaxis doses ranged from 25-50 IU/kg (for <12 years participants) and 20-40 IU/kg (for 12 years participants) with every-second-day treatment, or 25-60 IU/kg (for <12 years participants) and 20-50 IU/kg (for 12 years participants) with 3-times-weekly treatment. Bleeds and surgeries were treated in the same way as for the other two treatment groups (adolescents (13 to 16 years) and adults (17 and older)).
- Adolescents (13 to 16 Years); Adults (17 and Older): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. Participants who completed 6 months of treatment (prophylaxis or on-demand) in the main phase, were to continue the same treatment for up to approximately 18 months (extension phase). Participants were allowed to switch between treatments in the 'extension phase'. The recommended prophylaxis starting dose was 25 IU/kg. Prophylaxis doses ranged from 20-40 IU/kg (once every-second-day), or 20-50 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
Arm/Group | Older Children (8 to 12 Years) | Adolescents (13 to 16 Years) | Adults (17 and Older)
Number analyzed (Participants) | 22 | 6 | 18
Scores
  Baseline | 41.3 (16.4) | 42.2 (12.8) | 47.2 (13.8)
  Change from baseline: number analyzed (Participants) | 21 | 6 | 16
  Change from baseline | -10.1 (15.0) | -4.9 (8.8) | -6.3 (9.7)

39. Secondary Outcome: Change in Total Scores for Reported Health-related Quality of Life (for Parents): Month 6
Description: Reported results are baseline (month 0) and change from baseline (at month 6) of end of disease and age specific health related quality of life (HRQOL). HRQOL was collected through use of the PRO instrument, HAEMO-QOL (for parents of the children (4-7 years and 8-12 years)/adolescents (13-16 years)). HAEMO-QOL assessment included questions on physical health, feeling, view of himself, family, friends, perceived support, other persons, nursery School or Kindergarten, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Observed mean of the means of all the questions for HAEMO-QOL are presented.
Time Frame: Month 0, Month 6
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Scores
Groups:
- Small Children (4 to 7 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 30 IU/kg. Prophylaxis doses ranged from 25-50 IU/kg (once every-second-day), or 25-60 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
- Older Children (8 to 12 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. The recommended prophylaxis starting dose was 30 IU/kg (for <12 years participants) and 25 IU/kg (for 12 years participants). Prophylaxis doses ranged from 25-50 IU/kg (for <12 years participants) and 20-40 IU/kg (for 12 years participants) with every-second-day treatment, or 25-60 IU/kg (for <12 years participants) and 20-50 IU/kg (for 12 years participants) with 3-times-weekly treatment. Bleeds and surgeries were treated in the same way as for the other two treatment groups (small children (4 to 7 years) and adolescents (13 to 16 years)).
Arm/Group | Small Children (4 to 7 Years) | Older Children (8 to 12 Years) | Adolescents (12 to <18 Years)
Number analyzed (Participants) | 19 | 22 | 6
Scores
  Baseline: number analyzed (Participants) | 17 | 22 | 6
  Baseline | 45.7 (15.2) | 48.3 (14.1) | 40.8 (11.7)
  Change from baseline: number analyzed (Participants) | 18 | 22 | 6
  Change from baseline | -6.2 (7.7) | -9.9 (8.7) | -1.5 (7.2)

40. Secondary Outcome: Change in Total Scores for Reported Health-related Quality of Life (for Parents): Month 24
Description: Reported results are baseline (month 0) and change from baseline (at month 24) of end of disease and age specific health related quality of life (HRQOL). HRQOL was collected through use of the PRO instrument, HAEMO-QOL (for parents of the children (4-7 years and 8-12 years)/adolescents (13-16 years)). HAEMO-QOL assessment included questions on physical health, feeling, view of himself, family, friends, perceived support, other persons, nursery School or Kindergarten, sports and school, dealing with haemophilia, treatment, future, and relationships. Scores range for each question was 0-100, with a lower score indicating better quality of life related to haemophilia. Observed mean of the means of all the questions for HAEMO-QOL are presented.
Time Frame: Month 0, Month 24
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Scores
Groups:
- Small Children (4 to 7 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. Participants who completed 6 months of treatment (prophylaxis or on-demand) in the main phase, were to continue the same treatment for up to approximately 18 months (extension phase). Participants were allowed to switch between treatments in the 'extension phase'. The recommended prophylaxis starting dose was 30 IU/kg. Prophylaxis doses ranged from 25-50 IU/kg (once every-second-day), or 25-60 IU/kg (3-times-weekly). Bleeds were treated with one or more turoctocog alfa i.v. bolus injections as determined by the investigator and based on the WFH guidance. Participants who underwent surgery were treated with turoctocog alfa according to WFH guidance and their FVIII activity levels were to be maintained as per the following guidance: Minor surgery: 30-60 IU/dL. Major surgery: 80-100 IU/dL pre- and postoperatively.
- Older Children (8 to 12 Years): Participants were to receive turoctocog alfa i.v. injections for at least 6 months (main phase) as either prophylaxis or on-demand treatment at investigator's discretion. Participants who completed 6 months of treatment (prophylaxis or on-demand) in the main phase, were to continue the same treatment for up to approximately 18 months (extension phase). Participants were allowed to switch between treatments in the 'extension phase'. The recommended prophylaxis starting dose was 30 IU/kg (for <12 years participants) and 25 IU/kg (for 12 years participants). Prophylaxis doses ranged from 25-50 IU/kg (for <12 years participants) and 20-40 IU/kg (for 12 years participants) with every-second-day treatment, or 25-60 IU/kg (for <12 years participants) and 20-50 IU/kg (for 12 years participants) with 3-times-weekly treatment. Bleeds and surgeries were treated in the same way as for the other two treatment groups (small children (4 to 7 years) and adolescents (13 to 16 years)).
Arm/Group | Small Children (4 to 7 Years) | Older Children (8 to 12 Years) | Adolescents (13 to 16 Years)
Number analyzed (Participants) | 19 | 22 | 6
Scores
  Baseline: number analyzed (Participants) | 17 | 22 | 6
  Baseline | 45.7 (15.2) | 48.3 (14.1) | 40.8 (11.7)
  Change from baseline: number analyzed (Participants) | 19 | 21 | 6
  Change from baseline | -6.7 (11.5) | -11.3 (10.7) | -3.1 (3.9)

41. Secondary Outcome: Incremental Recovery of FVIII
Description: Blood samples for the evaluation of incremental recovery of FVIII were taken during a period of 48 hours post-dosing for participants 12 years and older and 24 hours post-dosing for participants below the age of 12 years. The incremental recovery was calculated as (FVIII: coagulant (C) activity measured in plasma 30 minutes after dosing - FVIII:C activity measured in plasma immediately before dosing)/(dose injected at time 0 minute), where the dose was expressed as IU FVIII product per kg body weight. The results are based on the chromogenic assay.
Time Frame: Days 1-2
Population: Full analysis set excluding outliers. The full analysis set included all dosed participants with data after dosing. Exceptional outlier pharmacokinetic (PK) profiles and/or individual plasma concentrations were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: (IU/mL)/(IU/kg BW)
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 4 | 6 | 3 | 4
(IU/mL)/(IU/kg BW) | 0.022 (0.003) | 0.026 (0.005) | 0.014 (0.007) | 0.026 (0.004)

42. Secondary Outcome: Area Under the Curve (AUC0-inf)
Description: Blood samples for the evaluation of AUC0-inf were taken during a period of 48 hours post-dosing for participants 12 years and older and 24 hours post-dosing for participants below the age of 12 years. AUC0-inf was defined as the area under the concentration versus time from time curve zero to infinity. The results are based on the chromogenic assay.
Time Frame: Days 1-2
Population: Full analysis set excluding outliers. The full analysis set included all dosed participants with data after dosing. Exceptional outlier PK profiles and/or individual plasma concentrations were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: IU*h/mL
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 3 | 6 | 3 | 4
IU*h/mL | 16.4 (3.5) | 17.7 (7.3) | 11.2 (4.7) | 16.9 (1.5)

43. Secondary Outcome: Half-life (t½)
Description: Blood samples for the evaluation of t½ were taken during a period of 48 hours post-dosing for participants 12 years and older and 24 hours post-dosing for participants below the age of 12 years. The results are based on the chromogenic assay.
Time Frame: Days 1-2
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 3 | 6 | 3 | 4
Hour (h) | 8.5 (1.4) | 8.3 (3.1) | 11.6 (0.6) | 8.4 (1.9)

44. Secondary Outcome: Clearance (CL)
Description: Blood samples for the evaluation of CL were taken during a period of 48 hours post-dosing for participants 12 years and older and 24 hours post-dosing for participants below the age of 12 years. The results are based on the chromogenic assay.
Time Frame: Days 1-2
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 3 | 6 | 3 | 4
mL/h/kg | 3.7 (0.9) | 3.5 (1.2) | 5.5 (2.2) | 3.5 (0.3)

45. Secondary Outcome: Highest Measured FVIII Activity in the Profile (Cmax)
Description: Blood samples for the evaluation of Cmax were taken during a period of 48 hours post-dosing for participants 12 years and older and 24 hours post-dosing for participants below the age of 12 years. The results are based on the chromogenic assay.
Time Frame: Days 1-2
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
Number analyzed (Participants) | 4 | 6 | 3 | 4
IU/mL | 1.2 (0.2) | 1.4 (0.3) | 0.9 (0.5) | 1.6 (0.2)

ADVERSE EVENTS:
Time Frame: All presented AEs are treatment emergent (TEAEs), which was defined as the events reported after trial product administration (day 1) until the end of the post-treatment follow-up period (i.e. month 24 + 14 days).
Description: The safety analysis set included participants who received at least one dose of the trial product.
Arm/Group | Small Children (0 to <6 Years) | Older Children (6 to <12 Years) | Adolescents (12 to <18 Years) | Adults (>=18 Years)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/33 | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/33 | 2/11 | 0/15
Other Adverse Events (participants affected / at risk) | 8/9 | 18/33 | 7/11 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Children (0 to <6 Years) (N=9) | Older Children (6 to <12 Years) (N=33) | Adolescents (12 to <18 Years) (N=11) | Adults (>=18 Years) (N=15)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Children (0 to <6 Years) (N=9) | Older Children (6 to <12 Years) (N=33) | Adolescents (12 to <18 Years) (N=11) | Adults (>=18 Years) (N=15)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Antiphospholipid antibodies positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (7) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puncture site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (7) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 2 (6) | 0 (0) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (12) | 7 (9) | 2 (3) | 3 (3)
Urethral disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mumps (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT02938585/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02938585/SAP_001.pdf